CLINICAL TRIAL: NCT01003002
Title: Determining the Natural History of Levodopa-Induced Dyskinesia (LID)
Brief Title: Natural History of Levodopa-Induced Dyskinesia (LID)
Status: Withdrawn | Type: Observational
Why Stopped: Funding not secured.
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Kathryn Chung, MD, Oregon Health & Science University
Other Study IDs: e4773
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2009-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Dyskinesia; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Movement Disorders | interventions — Levodopa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PD Cohort: The cohort for this study is Parkinson's disease patients that are beginning oral levodopa treatment within one month of the screening visit. This cohort has not previously (to the screening visit) been treated with oral levodopa.
  Interventions: Drug: Levodopa (delivered intravenously)

INTERVENTIONS:
Drug: Levodopa (delivered intravenously) — One mg/kg/hr of Levodopa will be given intravenously during inpatient testing days from 0900 to 1100.

SUMMARY:
Levodopa is the main drug treatment for Parkinson's disease. Levodopa can cause unwanted and uncontrolled movements called dyskinesias (LID). The severity of these movements can range from subtle to extremely debilitating. These movements may or may not interfere with normal activities such as putting on a coat or brushing ones teeth. Current estimates of the occurrence rate of LID range from 12 % to 100% after one year of levodopa treatment. These estimates used reporting mechanisms such as self-report and doctor-reported. These reporting mechanisms are not reliable. We will use an objective measure of dyskinesia in the first 5 years of treatment for Parkinson's disease. The purpose of this protocol is to use an objective measure to estimate dyskinesia onset.

DETAILED DESCRIPTION:
Nearly all Parkinson's disease (PD) patients eventually develop abnormal and unwanted movements (dyskinesias; LID) caused by the gold standard treatment, Levodopa. The severity of these movements can range from subtle to extremely debilitating and may or may not interfere with normal activities such as putting on a coat or brushing ones teeth. Current estimates of the prevalence of LID widely range from 12 % to 100% affected after one year. The purpose of this study is to estimate the median onset time of levodopa induced dyskinesia in newly treated Parkinson's disease patients. All participants will complete seven overnight visits at the OCTRI Inpatient unit over 5 years. During the next day, participants will complete a mental task while standing on a force plate for one minute every half hour until the end of the study. A levodopa IV infusion will occur from 0900 to 1100.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* At least 21 years of age
* Levodopa treatment that will be orally initiated no more than 1 month after the screening visit for the study.

Exclusion Criteria:

* Unable to stand for 1 minute intervals
* Sensory deficits in the feet
* Significant cognitive impairment
* Unstable medical or psychiatric conditions (including hallucinations)
* History of dopamine receptor blocking medications (Haldol, Orap, Zyprexa)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Levodopa-Induced Dyskinesia | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Chung, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Muller T, Woitalla D, Russ H, Hock K, Haeger DA. Prevalence and treatment strategies of dyskinesia in patients with Parkinson's disease. J Neural Transm (Vienna). 2007;114(8):1023-6. doi: 10.1007/s00702-007-0718-4. Epub 2007 Apr 10. PMID 17417738
- [Result] Parkinson Study Group. Pramipexole vs levodopa as initial treatment for Parkinson disease: A randomized controlled trial. Parkinson Study Group. JAMA. 2000 Oct 18;284(15):1931-8. doi: 10.1001/jama.284.15.1931. PMID 11035889
- [Result] Rascol O, Brooks DJ, Korczyn AD, De Deyn PP, Clarke CE, Lang AE. A five-year study of the incidence of dyskinesia in patients with early Parkinson's disease who were treated with ropinirole or levodopa. N Engl J Med. 2000 May 18;342(20):1484-91. doi: 10.1056/NEJM200005183422004. PMID 10816186
- [Result] Nutt JG, Carter JH, Lea ES, Sexton GJ. Evolution of the response to levodopa during the first 4 years of therapy. Ann Neurol. 2002 Jun;51(6):686-93. doi: 10.1002/ana.10189. PMID 12112073
- [Result] McColl CD, Reardon KA, Shiff M, Kempster PA. Motor response to levodopa and the evolution of motor fluctuations in the first decade of treatment of Parkinson's disease. Mov Disord. 2002 Nov;17(6):1227-34. doi: 10.1002/mds.10244. PMID 12465061